CLINICAL TRIAL: NCT00211900
Title: A Phase 3, Multicenter, Open-Label, Historical Comparative Study to Evaluate Immunogenicity and Safety of a Commercial Lot of StaphVAX®, a Bivalent Staphylococcus Aureus Glycoconjugate Vaccine in Adults on Hemodialysis
Brief Title: Evaluation of Manufacturing Lot of StaphVAX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nabi Biopharmaceuticals (Industry)
Responsible Party: Matt Hohenboken, MD, PhD, Executive Director, Clinical & Medical Affairs, Nabi Biopharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Nabi-1367
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-01-04 (Estimated); Status verified 2007-12

CONDITIONS: Staphylococcal Infections; Chronic Kidney Failure
MeSH Terms: conditions — Staphylococcal Infections; Kidney Failure, Chronic | interventions — StaphVax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vaccine (Experimental): single dose of StaphVAX in hemodialysis patients
  Interventions: Biological: S. aureus Type 5 & 8 Capsular Polysaccharide Vaccine

INTERVENTIONS:
Biological: S. aureus Type 5 & 8 Capsular Polysaccharide Vaccine — single IM dose totalling 200 mcg of conjugate
  Other Names: StaphVAX®

SUMMARY:
This study answers a U.S. Food and Drug Administration requirement for evaluation in people of a manufacturing lot of vaccine. Subjects receive one dose of one lot of vaccine. The antibodies in the blood measure the immunogenicity of the vaccine, and typical vaccine safety information is also collected.

ELIGIBILITY:
Inclusion Criteria:

* 8 wk of hemodialysis for ESRD,
* have written informed consent,
* a negative serum pregnancy test if appropriate,
* and expect to comply with protocol procedures and schedule

Exclusion Criteria:

* known HIV,
* immunomodulatory drugs,
* malignancy (other than basal cell or squamous cell carcinoma, carcinoma in situ of the cervix, or early stage prostate cancer),
* active infection in the 2 weeks prior to study injection,
* serious S. aureus infection within the last 3 months prior to injection,
* use of investigational drugs, vaccines or devices within the prior 30 days,
* hypersensitivity to components of StaphVAX

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-03; Primary Completion 2005-08 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Type-specific antibody concentrations | 6 weeks after vaccine dose

SECONDARY OUTCOMES:
Type-specific antibody concentrations | 3 weeks after vaccine dose
Elicited vaccine reactogenicity. | daily for 7 days after dose

CONTACTS AND LOCATIONS:
Overall Officials: Matt Hohenboken, MD, PhD, Study Director — Nabi Biopharmaceuticals
Locations (1):
- Trialogic Research, Madison, Alabama, United States